CLINICAL TRIAL: NCT05829070
Title: A Randomized Controlled Trial to Improve Health Insurance Literacy and Surveillance Among Young Adult Cancer Survivors
Brief Title: Improving Health Insurance Literacy Among Young Adult Cancer Survivors
Acronym: CHAT-S
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Intermountain Health (Unknown); Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Anne Kirchhoff, Associate Professor, Pediatrics, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R01CA276825 (NIH)
Record Dates: First submitted 2023-03-02; First posted 2023-04-25 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CHAT-S (Experimental): CHAT-S consists of 4 bi-weekly 35-45 minute videoconferencing sessions with a patient navigator and a patient booklet on insurance, costs, and survivorship care.
  Interventions: Behavioral: CHAT-S
- Usual Care (Placebo Comparator): Usual care will consist of a resource list sent by the navigator.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: CHAT-S — The CHAT-S intervention will include 4 videoconference sessions over a 2-month time period that is delivered by a patient navigator. Session 1 will include content to educate participants about survivorship care and common types of follow-up care required for their specific cancer, as well as, basic insurance terms and concepts. Session 2 will teach participants about their own insurance plan (e.g., coverage, benefits, breakdown of bills, and explanation of benefits) so they can better navigate both the medical and insurance systems. Session 3 reviews health insurance laws (e.g., ACA, FMLA, No Surprises Act) and how to proceed with an appeals process. Session 4 explains how to manage the costs through budgeting and cost-of-care conversations with their medical providers.
  Arms: CHAT-S
Behavioral: Usual Care — Usual care will consist of a resource list that describes organizational and community resources available on insurance, financial burden, and survivorship care. Further, we will track whether participants were referred or engaged in services using the follow-up surveys and via the EHR/claims data.
  Arms: Usual Care

SUMMARY:
We will conduct a randomized controlled trial to test a 4-session virtual health insurance navigation intervention that will increase knowledge about health insurance, reduce financial burden, and improve surveillance for recurrence among 300 young adult cancer survivors ages 26 to 39. We will combine self-reported survey data with electronic health records and claims data to examine the trial outcomes and efficacy. We will also conduct an economic evaluation using cost-effectiveness and budget impact analyses, to establish the sustainability of the intervention at improving outcomes of young adult survivors through increasing their health insurance knowledge and decreasing their financial burden.

DETAILED DESCRIPTION:
The first year after cancer treatment ends is a critical time to establish survivorship care for young adult (YA) cancer survivors ages 26 to 39. Receipt of evidence-based survivorship care, including surveillance for cancer recurrence based on national guidelines, remain low among YA survivors. At the same time, YAs ages 26 to 39 have the highest rate of both uninsurance and underinsurance among adults in the United States. Our team's prior work demonstrated that YA cancer survivors report low understanding of their health insurance and the services it covers, which affects their ability to navigate care. Together, these issues can lead to significant access to care barriers and severe medical cost consequences for this population. This proposal addresses the urgent need to improve YA cancer survivors' health insurance literacy and decrease financial toxicity, thus improving their ability to receive recommended survivorship care. Guided by Andersen and Aday's Behavioral Model of Health Services Use, we developed and pilot-tested a 4-session virtual patient navigation intervention for YA cancer survivors that was adapted from a pilot program for childhood cancer survivors. Initial results support feasibility, acceptability, and preliminary efficacy of both of these pilot trials with YA survivors ages 26 to 39. We now propose a randomized controlled trial to test the efficacy of this program ("CHAT-S," Cancer Health insurAnce Tools with Survivors) to improve health insurance literacy, financial toxicity due to medical costs, and post-treatment surveillance for recurrence among YA cancer survivors ages 26 to 39 (up to age 45). We plan to randomize N=300 (N=200 intervention; N=100 usual care) YAs with breast, testicular, lymphoma, sarcoma, and colorectal cancer who have completed initial treatment within the past year from 14 locations in the University of Utah Healthcare (UUHC) and Intermountain Healthcare (IH) systems. UUHC and IH have many rural (20%) and Hispanic/Latinx (18%) YA cancer survivors; we will oversample these important subgroups. We will determine whether CHAT-S improves health insurance literacy and financial toxicity at 6-month follow-up (primary outcomes). Further, UUHC and IH have an integrated data infrastructure which allows us to capture electronic health records and claims data to investigate whether CHAT-S improves surveillance care for recurrence at 18-month follow-up (secondary outcome). We will explore moderators (e.g., rurality, ethnicity) of the intervention effects. Finally, to inform future dissemination, we will conduct a budget impact analysis and a short-term and long-term time horizon cost-effectiveness analysis of CHAT-S. This proposal addresses the National Cancer Institute's goal of improving the care of cancer survivors and mitigating financial toxicity. We will demonstrate that a virtual health insurance literacy intervention can improve insurance literacy, financial toxicity, and surveillance care among YA cancer survivors, and provide guidance to improving survivorship care across the United States.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible for this study if they:

1. Were diagnosed with breast, testicular, lymphoma, sarcoma, and colorectal cancer,
2. Are between the ages of 26 to 45 years (preferably between 26-39, but no older than 45),
3. Have completed initial treatment (i.e., radiation, chemotherapy, or surgery) within the past year,
4. Are a patient at the University of Utah/Huntsman Cancer Institute or Intermountain Healthcare, and
5. Speak English.

Exclusion Criteria:

Potential participants will be excluded if they:

1. Are unable to participate due to developmental delay, and
2. Speak a language other than English, and
3. Unable to participate through either phone or a video capable computer or mobile device (e.g., smartphone, laptop, etc.).

Ages: 26 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2027-10 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Health Insurance Literacy Measure (HILM) | Baseline
  The degree to which individuals have the knowledge, ability, and confidence to find and evaluate information about health plans, select the best plan for their own (or their family's) financial and health circumstances, and use the plan. Determined by rating statements using a 4-point scale (very confident, somewhat confident, not too confident, not all confident).
COmprehensive Score for financial Toxicity (COST) | Baseline
  Financial distress related to medical costs. Determined by rating statements regarding financial distress on a 5-point scale (very much, quite a bit, somewhat, a little bit, not at all).
Health Insurance Literacy Measure | 6 months
  The degree to which individuals have the knowledge, ability, and confidence to find and evaluate information about health plans, select the best plan for their own (or their family's) financial and health circumstances, and use the plan. Determined by rating statements using a 4-point scale (very confident, somewhat confident, not too confident, not all confident).
COmprehensive Score for financial Toxicity (COST) | 6 months
  Financial distress related to medical costs. Determined by rating statements regarding financial distress on a 5-point scale (very much, quite a bit, somewhat, a little bit, not at all).
Health Insurance Literacy Measure | 12 months
  The degree to which individuals have the knowledge, ability, and confidence to find and evaluate information about health plans, select the best plan for their own (or their family's) financial and health circumstances, and use the plan. Determined by rating statements using a 4-point scale (very confident, somewhat confident, not too confident, not all confident).
COmprehensive Score for financial Toxicity (COST) | 12 months
  Financial distress related to medical costs. Determined by rating statements regarding financial distress on a 5-point scale (very much, quite a bit, somewhat, a little bit, not at all).

SECONDARY OUTCOMES:
Surveillance for Recurrence | 18 months
  Met (partly or fully) or failed to meet cancer surveillance for recurrence within the past year (looking from 6 months-18 months after baseline)
Survivorship Care Receipt | 18 months
  Gathering information regarding receiving other survivorship care (other than surveillance care) including shared, coordinated care (e.g., using current procedural terminology codes to designate having visits in the past year-6-18 months following baseline-with both primary care providers and oncologists).
Insurance Coverage | Baseline
  Questions asking about the type of insurance coverage participants have (having participants indicate if their coverage is public/private, policy holder, number of people covered etc).
Insurance Coverage | 6 months
  Questions asking about the type of insurance coverage participants have (having participants indicate if their coverage is public/private, policy holder, number of people covered etc).
Insurance Coverage | 12 months
  Questions asking about the type of insurance coverage participants have (having participants indicate if their coverage is public/private, policy holder, number of people covered etc).
Familiarity with the Affordable Care Act and other insurance legislation | Baseline
  Knowledge of protections (e.g., appeals), avenues for insurance coverage, and legal protections. Indicated using statements regarding familiarity with insurance legislation rated using a 4-point scale (very familiar, somewhat familiar, not too familiar, not at all familiar).
Familiarity with the Affordable Care Act and other insurance legislation | 6 months
  Knowledge of protections (e.g., appeals), avenues for insurance coverage, and legal protections. Indicated using statements regarding familiarity with insurance legislation rated using a 4-point scale (very familiar, somewhat familiar, not too familiar, not at all familiar).
Familiarity with the Affordable Care Act and other insurance legislation | 12 months
  Knowledge of protections (e.g., appeals), avenues for insurance coverage, and legal protections. Indicated using statements regarding familiarity with insurance legislation rated using a 4-point scale (very familiar, somewhat familiar, not too familiar, not at all familiar).
Feasibility of enrollment and session completion | 6 months
  Percentage enrolled calculated from number approached for participation and sessions completed calculated from total number enrolled in the intervention.
Acceptability: | 6 months
  5-point scales of satisfaction with CHAT-S. Rating statements regarding the study with a 5-point scale (very satisfied, somewhat satisfied, neutral, somewhat dissatisfied, very dissatisfied).
  assistance that you wanted? How helpful has this program been for you for accessing survivorship care?)
Patient Satisfaction with Interpersonal Relationship with Navigator | 6 months
  Experiences with communication and services provided by the navigator. Using statements from the Patient Satisfaction with Navigator Interpersonal Relationship (PSN-I). Using a 5-point scale (strongly agree, agree, neither agree nor disagree, disagree, strongly disagree).
Cost related literacy | Baseline
  Confidence in dealing with medical costs indicated by rating statements using a 4-point scale (very confident, somewhat confident, not too confident, not at all confident).
Cost related literacy | 6 months
  Confidence in dealing with medical costs indicated by rating statements using a 4-point scale (very confident, somewhat confident, not too confident, not at all confident).
Cost related literacy | 12 months
  Confidence in dealing with medical costs indicated by rating statements using a 4-point scale (very confident, somewhat confident, not too confident, not at all confident).

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided